CLINICAL TRIAL: NCT02936219
Title: Weaning of Preterm Infants During the First Year of Life: Impact on Anthropometry, Body Composition, Atopy and Neurodevelopmental Outcome
Brief Title: The PREWEAN Study. Weaning of Preterm Infants During the First Year of Life.
Acronym: PREWEAN
Status: Active, not recruiting | Type: Observational
Sponsor: Medical University of Vienna (Other)
Collaborators: Wilhelminenspital Vienna (Other); Kaiser Franz Josef Hospital (Other)
Responsible Party: Principal Investigator, Nadja Haiden,MD, Assoz. Prof. PD. Dr. Nadja Haiden, MSc, Medical University of Vienna
Other Study IDs: PREWEAN
Record Dates: First submitted 2016-10-14; First posted 2016-10-18 (Estimated); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Growth Failure; Atopy; Adiposity; Cognitive Impairment; Neurological Impairment
Keywords: complementary feeding; breast milk; formula feeding; combined feeding; preterm infants; body composition
MeSH Terms: conditions — Failure to Thrive; Obesity; Cognitive Dysfunction; Neurologic Manifestations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- Early complementary breast feeding: The EARLY complementary feeding group is defined as the introduction of complementary food <17th week of life corrected for term. In addition, infants are stratified to the milk regime, like human milk feeding, at the study enrollment.
- Early complementary combined feeding: The EARLY complementary feeding group is defined as the introduction of complementary food <17th week of life corrected for term. In addition, infants are stratified to the milk regime, like combined milk feeding, at the study enrollment.
- Early complementary formula feeding: The EARLY complementary feeding group is defined as the introduction of complementary food <17th week of life corrected for term. In addition, infants are stratified to the milk regime, like formula feeding, at the study enrollment.
- Late complementary breast feeding: The LATE complementary feeding group is defined as the introduction of complementary food ≥17th week of life corrected for term. In addition, infants are stratified to the milk regime, like human milk feeding, at the study enrollment.
- Late complementary combined feeding: The LATE complementary feeding group is defined as the introduction of complementary food ≥17th week of life corrected for term. In addition, infants are stratified to the milk regime, like combined milk feeding, at the study enrollment.
- Late complementary formula feeding: The LATE complementary feeding group is defined as the introduction of complementary food ≥17th week of life corrected for term. In addition, infants are stratified to the milk regime, like formula feeding, at the study enrollment.

SUMMARY:
In this Austrian observational study preterm infants born with a birth weight <1500 g and a gestational age <32 weeks will be investigated at the neonatal outpatient clinic. Infants will be stratified according their feeding regimen (breast, formula and combined feeding) and their introduction of solid foods (early complementary feeding group: <17th week of life corrected for prematurity, late complementary feeding group: ≥17th week of life corrected for prematurity). Nutrient intakes and anthropometric parameters will be assessed at term, 6 weeks, 12 weeks, 6 months, 9 months and 12 months - all corrected for prematurity and with 40, 54 and 66 months.

DETAILED DESCRIPTION:
Introduction: Evidenced-based guidelines for the introduction of complementary feeding in preterm infants are not available so far. In comparison to full-term babies, there is strong evidence that babies less than 1500 grams have increased nutritional needs starting with the time of birth up to the second year of life to establish catch up growth and to reach the main milestones in neurological development.

Evidence based data on feeding practices after discharge of the hospital, weaning and the quantity and quality of complementary food are missing. With this prospective observational study the investigators intend to close this knowledge gap in weaning of former preterm infants.

Methods: In this prospective observational study preterm infants born with a birth weight <1500 g and a gestational age <32 weeks will be recruited at term corrected for prematurity at the neonatal outpatient clinic. Infants will be stratified according their source of milk intake (breast milk, formula and mixed feeding) and their introduction of solid foods (early complementary feeding group: <17th week of life corrected for prematurity, late complementary feeding group: ≥17th week of life corrected for prematurity).

Nutritional intake will be estimated based on 24h Recalls at term and after 6 weeks of age corrected for prematurity. Furthermore, 3-days dietary records, an average dietary record and the introduction of the main food categories will be queried at 4 different time points (3 months, 6 months, 9 months and 12 months - all corrected for prematurity) by food questionnaire.

Within these visits anthropometric parameters (height, head circumference and weight), data on body composition (Pea Pod®, BodPod ) & bio-impedance measurements will be collected. Atopy will be determined by the clinical scoring system SCORAD. For follow up anthropometry and the neurodevelopmental outcome will be assessed by the Bayley Scale at 12 & 24 months corrected for prematurity and at 40 months of age. Furthermore, K-ABC II (Kaufmann assessment battery for children) will be performed at 66 months of age.

Goals: With this observational study the investigators aim to identify current feeding practices in premature infants and their impact on growth, body composition, atopy and neurodevelopmental outcome.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants born with a birth weight <1500g and a gestational age <32 weeks
* Informed consent

Exclusion Criteria:

* Gastrointestinal diseases: e.g. Hirschsprung disease
* Congenital heart diseases
* Major congenital birth defects
* Chromosomal aberrations

Ages: 1 Week to 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Preterm infants born with a birth weight <1500g and a gestational age <32 weeks
Sampling Method: Non-Probability Sample
Enrollment: 218 (Actual)
Dates: Start 2016-04; Primary Completion 2021-12 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Is there a height difference of 5% at one year of age corrected for prematurity between different complementary feeding groups? | The patients will be recruited in the period of 04/2016 till 06/2021. The primary observation period is one year.The follow up period lasts until 06/2025
  Is there a height difference of 5% at one year of age corrected for prematurity

SECONDARY OUTCOMES:
Atopy | 04/2016 till 06/2025
  Atopy measured by SCORAD
Body composition | 04/2016 till 06/2025
  Fat free mass measure by the body composition devices Peapod and Bodpod
Neurodevelopmental outcome with 1 and 2 years | 04/2017 till 06/2025
  Neurodevelopmental outcome measured by the Bailey III with 1 and 2 years of age corrected for prematurity
Neurodevelopmental outcome with 4,5 and 5,5 years | 04/2017 till 06/2025
  Neurodevelopmental outcome measured with the KABC- II by 54 and 66 moths of age
weight | 04/2016-06/2025
  weight in g or kg
head circumference | 04/2016-06/2025
  in cm

CONTACTS AND LOCATIONS:
Overall Officials: Nadja Haiden, Principal Investigator — Medical University of Vienna, 1090 Vienna, Austria
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided